CLINICAL TRIAL: NCT00546117
Title: A Clinical Trial of Proton Pump Inhibitors to Treat Children With Chronic Otitis Media With Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Doris Duke Charitable Foundation (Other); TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Principal Investigator, Judith Lieu, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRPO# 07-0762
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Otitis Media With Effusion
Keywords: otitis media with effusion; gastroesophageal reflux; ear infection; proton pump inhibitor
MeSH Terms: conditions — Otitis Media with Effusion; Gastroesophageal Reflux; Otitis | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lansoprazole (Prevacid) (Experimental): Prevacid SoluTab (15 or 30 mg tab) once daily for 2 months
  Interventions: Drug: lansoprazole
- Placebo (Placebo Comparator): Placebo SoluTab once daily for 2 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lansoprazole — Prevacid SoluTab 15 mg daily by mouth for 2 months (patients weighing 10-30 kg),or Prevacid SoluTab 30 mg daily by mouth for 2 months (patients weighing >30 kg) is the experimental arm. Placebo Solutabs will be given in the same dosage, frequency, and duration for the placebo arm.
  Other Names: Prevacid SoluTab
  Arms: Lansoprazole (Prevacid)
Drug: placebo — Placebo Solutab in 15 and 30 mg dosages.
  Other Names: Placebo Solutab
  Arms: Placebo

SUMMARY:
This study is being done to see if reflux of stomach fluid might be a cause of chronic fluid in the ears. Our hypothesis is that treatment with an anti-reflux medication (lansoprazole) will increase the rate of resolution of chronic middle ear fluid in children.

DETAILED DESCRIPTION:
This study is being done to see if reflux of stomach fluid might be a cause of fluid in the ears. Earlier studies have found pepsin or pepsinogen, a component of stomach fluid, in the middle ear fluid of many children with chronic middle ear fluid. Anti-reflux medicines called proton pump inhibitors (PPI) reduce the acidity of the contents of the stomach and the activity of pepsin or pepsinogen. We are studying the effectiveness of a PPI called lansoprazole (Prevacid™) in reducing fluid in the ears. If lansoprazole is able to reduce the fluid in the middle ear, this tells us that the reflux of gastric acid into the esophagus and into the ear canal may be causing middle ear fluid.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic otitis media with effusion meeting clinical indications for tympanostomy tubes placement, defined as the presence of middle ear fluid on physical exam for at least 3 months, in at least one ear.

Exclusion Criteria:

* Past medical history or concurrent conditions known to increase the incidence of either recurrent otitis media or otitis media with effusion or gastroesophageal reflux disease, including cleft palate, neurological delay, cerebral palsy, Down syndrome, velocardiofacial syndrome, and primary ciliary dyskinesia.
* Children with structural abnormalities of the tympanic membranes, such as cholesteatoma, deep retraction pockets, and atelectasis of the tympanic membrane. These abnormalities would require placement of tympanostomy tubes in standard clinical practice.
* Children weighing less than 10 kilograms, due to the lower weight limit for standard Prevacid™ dosing

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith EC Lieu, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Lieu JE, Muthappan PG, Uppaluri R. Association of reflux with otitis media in children. Otolaryngol Head Neck Surg. 2005 Sep;133(3):357-61. doi: 10.1016/j.otohns.2005.05.654. PMID 16143181
- [Background] Tasker A, Dettmar PW, Panetti M, Koufman JA, P Birchall J, Pearson JP. Is gastric reflux a cause of otitis media with effusion in children? Laryngoscope. 2002 Nov;112(11):1930-4. doi: 10.1097/00005537-200211000-00004. PMID 12439157
- [Background] Abd El-Fattah AM, Abdul Maksoud GA, Ramadan AS, Abdalla AF, Abdel Aziz MM. Pepsin assay: a marker for reflux in pediatric glue ear. Otolaryngol Head Neck Surg. 2007 Mar;136(3):464-70. doi: 10.1016/j.otohns.2006.08.030. PMID 17321879
- [Background] Sone M, Yamamuro Y, Hayashi H, Yanagi E, Niwa Y, Nakashima T. Prediction of gastroesophageal reflux in otitis media with effusion in adults. Acta Otolaryngol. 2007 May;127(5):470-3. doi: 10.1080/00016480600868406. PMID 17453471

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevacid: Prevacid SoluTab (15 or 30 mg tab) once daily for 2 months
Period: Overall Study
Arm/Group | Prevacid | Placebo
Started | 9 | 7
Completed | 5 | 7
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Inability to schedule follow-up visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevacid | Placebo | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 7 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.82 (1.98) | 5.45 (1.32) | 5.10 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Absence of Middle Ear Fluid by Pneumatic Otoscopy, Right Ear
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Prevacid | Placebo
Number analyzed (Participants) | 9 | 7
participants | 1 | 0

2. Primary Outcome: Absence of Middle Ear Fluid by Pneumatic Otoscopy, LeftEar
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Prevacid | Placebo
Number analyzed (Participants) | 9 | 7
participants | 1 | 3

3. Secondary Outcome: Acoustic Reflectometry: Level of Risk as Defined by Manufacturer
Description: Spectral gradient acoustic reflectometry is a noninvasive, non-audible acoustic wave used to help detect middle ear fluid. The manufacturer recommends interpretation of the angle result as: <49°, high risk of middle ear effusion (level 5); 49-59°, moderate-high risk (level 4); 60-69°, moderate risk (level 3); 70-95°, low-moderate risk (level 2) and >95°, low risk (level 1).
Time Frame: 2 months
Measure: Mean (Full Range); unit: level of risk
Arm/Group | Lansoprazole (Prevacid) | Placebo
Number analyzed (Participants) | 9 | 7
level of risk | 2.5 [1 to 5] | 3.5 [1 to 5]

4. Secondary Outcome: Number of Participants With Normal Type A Tympanometry
Description: Tympanometry of both ears, coded by Jerger classification (Type A, normal; type B, flat; Type C; negative pressure).
  This is a standard test of middle ear status as performed by audiologists. Please refer to the reference for more information: Kileny & Zwolan, Diagnostic Audiology, chapter 133, Cummings Otolaryngology-Head and Neck Surgery, Elsevier/Saunders, 2015.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lansoprazole (Prevacid) | Placebo
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With at Least 1 Symptoms of Reflux in the Past Week, Assessed by the Reflux Symptom Questionnaire
Description: Questions regarding reflux symptoms, created and evaluated by Nelson et al, Prevalence of symptoms of gastroesophageal reflux during childhood: a pediatric practice-based survey, Arch Pediatr Adolesc Med 2000;154;150-154. This study used the GER3-9P version for children aged 3-9 years. Results are reported as number reporting at least one specific symptom in the past week, maximum 7 symptoms.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lansoprazole (Prevacid) | Placebo
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Prevacid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No